CLINICAL TRIAL: NCT04292236
Title: The Effect of Food Supplements on Food Intake and Gut Hormone Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: QMREC2018/20
Record Dates: First submitted 2020-02-20; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Obesity; Endocrine; Obesity; Appetite; Perverted
Keywords: Nutrient; Anorexigenic hormone; Calorific Intake
MeSH Terms: conditions — Obesity | interventions — lauric acid; perilla seed oil; 3,3'-diindolylmethane

STUDY DESIGN:
Intervention Model Description: Double blinded, randomised, crossover, placebo controlled.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Administered at time 0 min and 300 min. Cellulose was used as the placebo.
  Interventions: Dietary Supplement: Lauric Acid, Perilla Oil and Diindolylmethane
- Dietary Supplement (Active Comparator): Administered at 0 min and 300 min. Combination of lauric acid, perilla oil and diindolylmethane was used as the dietary supplement.
  Interventions: Dietary Supplement: Lauric Acid, Perilla Oil and Diindolylmethane

INTERVENTIONS:
Dietary Supplement: Lauric Acid, Perilla Oil and Diindolylmethane — Colonic release capsules containing lauric acid (2400mg), perilla oil (2100mg) and diinodlylmethane (500mg) given to volunteers 1 hour prior to standardised breakfast and lunch meal. Placebo group given cellulose capsules of same volume prior to standardised breakfast and lunch meal.

SUMMARY:
When a meal is eaten, nutrients activate the release of hormones from the bowel into the blood stream. Normally there is a large amount of hormone released, which tells the brain that an individual is full and to stop eating. When people gain weight and become overweight or obese, these hormone signals are reduced, resulting in these people eating more and gaining more weight. This study is investigating mechanisms which may break this cycle by using particular nutrients to restore reduced hormone levels.

ELIGIBILITY:
Inclusion Criteria:

* Obese but otherwise healthy volunteers,
* body mass index (BMI) of 30-40 kg/m2
* agreement to consume scheduled meals
* ability to understand the study information sheet and instructions in English and able to provide informed consent.

Exclusion Criteria:

* Not meeting any of the exclusion criteria above.
* Major gut surgery
* Major health problems
* Taking medication for diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Effect on appetite and satiety ratings | Study day 1 and study day 2 (following meal intake at breakfast and lunch)
  Effect on appetite measured as change in calorific intake

SECONDARY OUTCOMES:
Effect on gut hormone levels | Study day 1 and study day 2 with samples taken every 30 min
  Assess changes to circulating levels of anorectic hormones GLP-1, PYY and orexigenic hormone Ghrelin.
Effect on satiety scores | Study day 1 and study day 2 (following meal intake at breakfast and lunch)
  Using a visual analogue scale measuring changes to hunger, satiety and fullness scores

CONTACTS AND LOCATIONS:
Overall Officials: Madusha Peiris, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Queen Mary University of Queensland, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peiris M, Aktar R, Reed D, Cibert-Goton V, Zdanaviciene A, Halder W, Robinow A, Corke S, Dogra H, Knowles CH, Blackshaw A. Decoy bypass for appetite suppression in obese adults: role of synergistic nutrient sensing receptors GPR84 and FFAR4 on colonic endocrine cells. Gut. 2022 May;71(5):928-937. doi: 10.1136/gutjnl-2020-323219. Epub 2021 Jun 3. PMID 34083384